CLINICAL TRIAL: NCT06473727
Title: Evaluation of the Initial Color Match of Anterior Non-caries Cervical Lesions Restorated With Different Single-shade Resin Composites: A Randomized Clinical Study
Brief Title: Evaluation of the Initial Color Match of Different Single-shade Composites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ayse Nur Dogan, Lecturer, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ErciyesU-DF-AD-01
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Dental Diseases
Keywords: blending; color match; composite resin; esthetics
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Intervention Model Description: Two groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omnichoroma (Active Comparator): Anterior non-carious cervical lesions restored with Omnichoroma single-shade resin composite.
  Interventions: Other: Omnichoroma
- Charisma Topaz One (Active Comparator): Anterior non-carious cervical lesions restored with Charisma Topaz One single-shade resin composite.
  Interventions: Other: Charisma Topaz One

INTERVENTIONS:
Other: Omnichoroma — Patients with anterior non-carious cervical lesions were treated with Omnichoroma. Colour measurements were taken from the middle third of the teeth to be treated using a spectrophotometer. The initial colour measurement was taken from the middle third of the restoration made in the same place and at the same time 24 hours after treatment.
  Other Names: Group 1
  Arms: Omnichoroma
Other: Charisma Topaz One — Patients with anterior non-carious cervical lesions were treated with Charisma Topaz One. Colour measurements were taken from the middle third of the teeth to be treated using a spectrophotometer. The initial colour measurement was taken from the middle third of the restoration made in the same place and at the same time 24 hours after treatment.
  Other Names: Group 2
  Arms: Charisma Topaz One

SUMMARY:
The aim of this study was to evaluate the initial colour match of anterior non-carious cervical lesions restored with different single-shade resin composites, namely Omnichroma (Tokuyama) and Charisma Topaz One (Kulzer).

DETAILED DESCRIPTION:
Colour selection for composite restorations is a challenging process influenced by a number of environmental and operator factors. The polychromatic structure of natural teeth presents a challenge to shade selection. Consequently, the prevailing trend towards simplification of shade matching has led to the emergence of single-shade universal composites. Single-shade universal composites are able to replicate the natural colour of teeth by capturing the structural colour based on the size of the filler particles. Unlike other materials, it does not require the use of additional dyes or pigments. The blending, colour induction and colour assimilation effects of resin composites are collectively referred to as the chameleon effect. This phenomenon allows resin-based restorative materials to achieve a shade that closely resembles the colour of the surrounding tooth structure. The intelligent monochromatic composite makes shade selection easier for the clinician and provides a quick and easy way to create aesthetic restorations. Its distinctive character reduces confusion and potentially saves time in the clinic. However, the effectiveness of this material in matching different shades of natural teeth remains uncertain, and there is a paucity of clinical evidence on the efficacy of its colour-matching capabilities in dental restorations.

ELIGIBILITY:
Inclusion Criteria:

* Maintain satisfactory oral hygiene
* Have healthy gingival tissues
* Presence of an anterior non-carious cervical lesion approximately 5 m wide

Exclusion Criteria:

* Presence of caries
* Signs of fistula
* Pulp exposure
* Periodontal tissue swelling
* Abnormal tooth mobility

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-06-16 (Actual)

PRIMARY OUTCOMES:
Color assesment | 24 hours
  The color match of all restorations was evaluated with a spectrophotometer.The values of the coordinates L*, a* and b* in the middle third of the tooth before the restorations and after 24 hours in the middle third of the restorations were evaluated using a digital spectrophotometer. The colour difference (ΔE00) was calculated using an Excel spreadsheet with parametric factors set to 1.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Nur Dogan, Principal Investigator — TC Erciyes University
Locations (1):
- Faculty of Dentistry, Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No